CLINICAL TRIAL: NCT07179848
Title: Phase I Clinical Trial of a New Non-invasive Deep Brain Stimulation Technique
Brief Title: Safety and Feasibility of Temporal Interference Brain Stimulation for Treatment in Psychiatric Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-04-001A; NSTC 112-2321-B-A49-013 (Other Grant/Funding Number: National Science and Technology Council (NSTC))
Record Dates: First submitted 2025-08-28; First posted 2025-09-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Health Adults; Temporal Interference Stimulation; Safety and Effectiveness; Crossover Study
Keywords: Hippocampus; Temporal Interference Stimulation; Insula; Anterior Cingulate Cortex; Inferior Frontal Cortex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Hippocampus - Treatment first (Experimental)
  Interventions: Device: Temporal Interference Stimulation - Treatment first
- Hippocampus - Sham first (Sham Comparator)
  Interventions: Device: Temporal Interference Stimulation - Sham first
- Insula - Treatment first (Experimental)
  Interventions: Device: Temporal Interference Stimulation - Treatment first
- Insula - Sham first (Sham Comparator)
  Interventions: Device: Temporal Interference Stimulation - Sham first
- Anterior cingulate cortex - Treatment first (Experimental)
  Interventions: Device: Temporal Interference Stimulation - Treatment first
- Anterior cingulate cortex - Sham first (Sham Comparator)
  Interventions: Device: Temporal Interference Stimulation - Sham first
- Inferior frontal cortex - Treatment first (Experimental)
  Interventions: Device: Temporal Interference Stimulation - Treatment first
- Inferior frontal cortex - Sham first (Sham Comparator)
  Interventions: Device: Temporal Interference Stimulation - Sham first

INTERVENTIONS:
Device: Temporal Interference Stimulation - Treatment first — Receive treatment stimulation for 5 consecutive days, followed by a 2-days washout period, then complete the remaining 5 days of sham stimulation
  Arms: Anterior cingulate cortex - Treatment first; Hippocampus - Treatment first; Inferior frontal cortex - Treatment first; Insula - Treatment first
Device: Temporal Interference Stimulation - Sham first — Receive sham stimulation for 5 consecutive days, followed by a 2-days washout period, then undergo 5 days of treatment stimulation
  Arms: Anterior cingulate cortex - Sham first; Hippocampus - Sham first; Inferior frontal cortex - Sham first; Insula - Sham first

SUMMARY:
The goal of this clinical trial is to validate if temporal interference brain stimulation (TIBS) is safe in healthy volunteers aged 20 to 65. The main questions it aims to answer are:

* Is it safe to apply TIBS intervention to the left hippocampus in healthy participants?
* Is it safe to apply TIBS intervention to the left insula in healthy participants?
* Is it safe to apply TIBS intervention to the left anterior cingulate cortex in healthy participants?
* Is it safe to apply TIBS intervention to the right inferior frontal cortex in healthy participants?

Participants will:

* Be Randomly allocated to either sham-first group or treat first-group, stratified by stimulated brain region, following a crossover-controlled experimental design
* Complete baseline cognitive evaluations and mental status assessments, and undergo a baseline MRI scan on the same day
* Receive stimulation for 5 consecutive days, followed by a 2-days washout period, then complete the remaining 5 days of stimulation.
* Complete post-intervention cognitive evaluations and mental status assessments, and undergo a post-intervention MRI scan on the same day

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults from the community
* Age between 20 and 65 years old
* No diagnosis of severe psychiatric disorders
* No family history of psychiatric diseases

Exclusion Criteria:

* Age below 20 years old or above 65 years old
* Currently prescribed any medication
* Diagnosis of psychiatric disorders (e.g., Major Depressive Disorder, Bipolar Disorder, Schizophrenia)
* Diagnosis of neurological disorders (e.g., Dementia, Stroke, Parkinson's disease)
* History of substance abuse
* Diagnosis of cancer or malignant tumors
* Chronic kidney failure or undergoing hemodialysis
* Pregnant or breastfeeding
* Severe arrythmia, presence of pacemaker, or metal implants in the brain
* Claustrophobia
* History or family history of seizure
* History of syncope
* Organic brian disease, brian trauma, or history of neurosurgery
* Received electroconvulsive therapy or repetitive transcranial magnetic stimulation within the past month
* Skin disorders (e.g., dermatitis, psoriasis, eczema)
* Currently participating in other clinical interventional trials
* Presence of any metal implants or devices affected by electromagnetic fields

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Changes in NRS related to intervention | Baseline (before each stimulation session), midpoint during each session, immediately after each stimulation for 10 sessions (approximately 2 weeks), and 1 month after completion of all sessions.
  Numeric rating scale (NRS) will be used to evaluate the side effects, pain intensity, and other adverse events potentially related to the intervention, at baseline, during stimulation, immediately after each session, and at follow-up.
Changes in VAS related to intervention | Baseline (before each stimulation session), midpoint during each session, immediately after each stimulation for 10 sessions (approximately 2 weeks), and 1 month after completion of all sessions.
  Visual analog scale (VAS) will be used to evaluate the side effects, pain intensity, and other adverse events potentially related to the intervention, at baseline, during stimulation, immediately after each session, and at follow-up.
Changes in MMSE from baseline to post-intervention | Approximately 1 week prior to the first stimulation session and approximately 1 week following the last stimulation session
  Mini-Mental State Examination (MMSE) will be administered to evaluate cognitive function approximately 1 week before the first intervention and 1 week after the last intervention. Cognitive function will be considered normal if the MMSE score is greater than 24.
Changes in BAI from baseline to post-intervention | Approximately 1 week prior to the first stimulation session and approximately 1 week following the last stimulation
  Beck Anxiety Inventory (BAI) will be administered to evaluate the mental status approximately 1 week before the first intervention and 1 week after the last intervention. Mental status will be considered stable if both BAI and BDI are less than 13.
Changes in BDI from baseline to post-intervention | Approximately 1 week prior to the first stimulation session and approximately 1 week following the last stimulation
  Beck Depression Inventory (BDI) will be administered to evaluate the mental status approximately 1 week before the first intervention and 1 week after the last intervention. Mental status will be considered stable if both BAI and BDI are less than 13.
Changes in MRI from baseline to post-intervention | Approximately 1 week prior to the first stimulation session and approximately 1 week following the last stimulation
  T1-weighted magnetic resonance imaging (T1-weighted MRI) and resting-state functional magnetic resonance imaging (resting-state fMRI) will be acquired to evaluate structural and functional brain alterations potentially related to the intervention. Imaging will be performed approximately 1 week before the first intervention and 1 week after the last intervention.

SECONDARY OUTCOMES:
Changes in WCST score from baseline to post-intervention | Approximately 1 week prior to the first stimulation session and approximately 1 week following the last stimulation session
  Wisconsin Card Sorting Test (WCST) will be administered to evaluate cognitive function approximately 1 week before the first intervention and 1 week after the last intervention.
Changes in verbal fluency test from baseline to post-intervention | Approximately 1 week prior to the first stimulation session and approximately 1 week following the last stimulation session
  Verbal fluency test will be administered to evaluate cognitive function approximately 1 week before the first intervention and 1 week after the last intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Due to the limited sample size, the risk of participant re-identification may be higher.